CLINICAL TRIAL: NCT04620629
Title: The Effect of Probiotic Supplement on Urinary D-lactic Acid Level in Newborns Receiving Antibiotic Treatment
Brief Title: The Effect of Probiotic Supplement on Urinary D-lactic Acid Level in Newborns
Status: Completed | Type: Observational
Sponsor: H. Tolga Çelik (Other)
Responsible Party: Sponsor-Investigator, H. Tolga Çelik, Principal Investigator, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: KA-19134
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Antibiotic Side Effect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: Late premature and term babies without any disease
- probiotic group: Babies whose probiotic support is started and continues because they cannot receive breast milk, and whose antibiotic treatment is started in the neonatal period.
- antibiotic group: Babies who receives antibiotic treatment in the neonatal period and does not receive probiotic support before.

SUMMARY:
It is thought that prophylactic enteral probiotics in newborns may play a role in the prevention of infection and NEC-related morbidity by preventing bacterial migration in the mucosa, reducing their number by competing with pathogenic bacteria, providing microbial balance, and increasing intestinal immunity.

In our study, it was determined to detect normal D-lactic acid levels in urine in late premature (babies born after 34 weeks of gestation) and term babies, to show the negative effect of antibiotic treatment on the intestinal flora indirectly by measuring urinary D-lactic acid, and the probiotic support in babies using antibiotics was disrupted. The investigators aim to investigate hypothesis that it will have a corrective effect on the intestinal flora by comparing urinary D-lactic acid levels.

DETAILED DESCRIPTION:
Lactic acid exists as two optical isomers, L-lactic acid and D-lactic acid. These isomers are metabolized to or synthesized from pyruvate by the action of isomer-specific enzymes (L-lactate dehydrogenase and D-lactate dehydrogenase). Mammals, including humans, do not possess D-lactate dehydrogenase, and therefore D-lactate production in human tissue is very limited. The endogenous single D-lactate synthesis known in man is carried out by glyoxalase. In this pathway, methylglyoxal is converted into D-lactate by the enzymes glyoxalase-1 and glyoxalase-2. Due to this restricted production, the blood D-lactate level in healthy people is so low that L-lactate is the major physiological enantiomer of lactate in the human body.

The bacterial flora in the human gastrointestinal tract has the ability to produce L and / or D-lactate depending on the amount of L-LDH and D-LDH present. Some strains of bacteria have the enzyme DL-lactate racemase to convert one isomer to another. Therefore, racemization reactions can further increase the amount of D-lactate isomers present in the column. Although there is no D-lactate dehydrogenase enzyme in humans, D-Lactate is metabolized into pyruvate by the enzyme D-2-hydroxy acid dehydrogenase (D-2-HDH), an intramitochondrial flavoprotein with high activity in the liver and renal cortex. The kidney's threshold for D-lactate is much lower than L-lactate and is efficiently excreted in urine as well as metabolic clearance. Thus, under normal conditions, D-lactate produced by tissue metabolism or bacterial fermentation in the gut; It does not cause a clinically significant increase in lactate in blood, urine or feces.

D-lactic acidosis is a well-defined complication of short bowel syndrome due to the combination of altered gastrointestinal tract anatomy and abnormal bacterial flora. Many case reports reported in the literature are associated with short bowel syndrome secondary to various causes. There are studies investigating the effects of fermented formulas and probiotics on D-lactic acid in healthy babies. In these studies, no increased risk for D-lactic acidosis was found in healthy infants fed with probiotic supplemented formulas.

Considering the studies on newborns; In babies with necrotizing enterocolit, it has been shown that urinary D-lactate excretion increased as a result of increased enteric bacterial activity. In another study, plasma D-lactic acid level was found to be high in premature babies with necrotizing enterocolitis. However, more detailed studies on newborns are needed.

ELIGIBILITY:
Inclusion Criteria:

* Late preterm and term babies
* Babies who are fed only breast milk and / or formula with breast milk
* Babies who have to be given formula support in the early period because they cannot receive breast milk or are not sufficient in the neonatal period, therefore probiotic support is started and continues
* Babies whose antibiotic treatment is started in the neonatal period
* Babies whose parents consent to participate in the study

Exclusion Criteria:

* Hypoxic ischemic encephalopathy
* Babies with urinary tract infections
* Babies with a history of premature rupture of membranes
* Chromosomal abnormality
* Those with major congenital anomaly, gastrointestinal system anomaly
* Presence of any known immunodeficiency,

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy newborns who born after 34 weeks of gestation, late preterm and term infants receiving antibiotic treatment,
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
urinary D-lactate levels | 4 weeks
  Urinary D-lactic acid levels of infants in the subgroup taking probiotics and not taking probiotics will be compared at the end of the 4th week.

CONTACTS AND LOCATIONS:
Overall Officials: Tolga Celik, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)